CLINICAL TRIAL: NCT06159075
Title: Reducing Self-Stigma Among Individuals with History of Childhood Maltreatment: a Cross-Cultural Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Yuval Y Neria, Professor, and Director of PTSD at Columbia University, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 8453a
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Stigma, Social; Child Abuse; Child Neglect; Help-Seeking Behavior
MeSH Terms: conditions — Social Stigma; Help-Seeking Behavior | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Video with Childhood Maltreatment-Related Content (Experimental): Participants will view a video of an actor describing the story of an individual who experienced childhood maltreatment and how they overcame its effects on their life.
  Interventions: Behavioral: Video
- Control Video (No Intervention): Participants in this arm will view a same-length video with the same actor, but without a personal narrative of CM experience.

INTERVENTIONS:
Behavioral: Video — A short video aimed at reducing self-stigma among individuals with a history of childhood maltreatment and increasing their help seeking intentions (if needed).
  Arms: Video with Childhood Maltreatment-Related Content

SUMMARY:
Individuals who report experiencing any kind of abuse during childhood report shame and self-blame, often leading to self-stigma and a reluctance to reveal their experiences and seek help. Such stigma may aggravate the mental health consequences of child maltreatment (CM).

The investigators hypothesize that:

1. The brief video-based intervention will have the immediate and repeated effect of reducing self-stigma among CM survivors compared with the control condition.
2. The brief video-based intervention will increase seeking treatment compared with the control condition.
3. The brief video-based intervention will show similar effects in reducing self-stigma across multiple countries.

DETAILED DESCRIPTION:
Prior research suggests that social contact-based interventions are the most efficient way of reducing stigma. This study aims to address self-stigma and empower individuals who self-reported experiencing any kind of abuse during childhood and increase their openness to seeking help, if needed.

Four hundred participants with self-reported experience of any kind of childhood abuse will be recruited to participate in a Randomized Controlled Trial (RCT) testing the efficacy of the intervention. Participants will be randomized into one of two arms: 1) A 2-minute video intervention in which a CM survivor (presented by an actor) shares their personal CM experience and describes how they were able to overcome feelings of shame and self-blame to seek mental health care; or 2) A 2-minute control video using the same actor, but without a personal narrative of CM experience. Both videos will be preceded by and immediately followed by questionnaires assessing self-stigma and openness to seeking treatment. An additional assessment of emotional engagement will be added immediately following intervention delivery. Following the intervention, there will be a 30- day follow-up to examine potential long-term effects.

The results will be analyzed alongside results from parallel protocols being conducted by partner sites in other countries (Switzerland, Sweden, Japan, Peru, India, Australia, Turkey, South Africa, and Israel). Each site will conduct the study under their own university's purview and with their own protocol, and only deidentified data will be shared for analysis.

All study procedures will be conducted remotely via CloudReseach and Mechanical Turk, which is a crowdsourcing platform. The study survey will be hosted by Qualtrics.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* US resident
* Individuals who endorse yes to one of the following items: physical aggression in family or household, emotional or verbal abuse in family or household, sexual abuse or inappropriate sexual experiences, negligence - physical or emotional, mental illness or substance abuse at home, incarceration of family member
* Fluent in English and able to give informed consent

Exclusion Criteria:

- N/A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 964 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Self-Stigma Questionnaire - Post-Intervention | Immediately post-intervention
  Change in stigma items from baseline - higher score indicates higher stigma (range of 15 to 60)
Self-Stigma Questionnaire - Follow-Up | 30 days post-intervention
  Change in stigma items from baseline - higher score indicates higher stigma (range of 15 to 60)
Help Seeking Intentions - Post-Intervention | Immediately post-intervention
  Change in treatment-seeking intentions from baseline - higher score indicates higher help-seeking intentions (range of 3 to 12)
Help Seeking Intentions - Follow-Up | 30 days post-intervention
  Change in treatment-seeking intentions from baseline - higher score indicates higher help-seeking intentions (range of 3 to 12)

CONTACTS AND LOCATIONS:
Overall Officials: Yuval Neria, PhD, Principal Investigator — NYSPI and Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No